CLINICAL TRIAL: NCT02848807
Title: Chemotherapy-related Toxicity, Nutritional Status and Quality of Life in Precachectic Oncologic Patients With or Without High Protein Nutritional Support. A Prospective, Randomized Study
Brief Title: Chemotherapy-related Toxicity, Nutritional Status and Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Clinical Centre, Gdansk (Other)
Collaborators: Nutricia Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 01/2014/UCK
Record Dates: First submitted 2014-07-16; First posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Toxicity Due to Chemotherapy; Cancer Cachexia; Metastatic Colorectal Cancer; Quality of Life; Dietary Modification
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Dietary Supplements

ARMS (2):
- NUTRIDRINK Compact Protein (Active Comparator): NUTRIDRINK Compact Protein Oral nutritional supplement Dietary advice
  Interventions: Dietary Supplement: NUTRIDRINK Compact Protein
- without oral nutritional supplements (No Intervention): Dietary advice alone

INTERVENTIONS:
Dietary Supplement: NUTRIDRINK Compact Protein — high-energy, high-protein, oral liquid nutritional supplement; dosage: 2x125 ml per day, 7 days per week for 12 weeks (3 months)
  Other Names: Oral nutritional supplement
  Arms: NUTRIDRINK Compact Protein

SUMMARY:
Determine whether nutritional support with high protein ONS in adult oncologic patients in the first step of cancer cachexia - asymptomatic precachexia, influence on the toxicity of systemic therapy.

DETAILED DESCRIPTION:
Other endpoints:

* to determine whether high protein ONS influence on the nutritional status
* to determine whether high protein ONS influence on the quality of life
* to determine whether high protein ONS influence on the performance status
* to determine high protein ONS tolerability / ONS intake compliance

ELIGIBILITY:
Inclusion Criteria:

* histological confirmed diagnosis of CRC in clinical stage IV
* successful qualification to chemotherapy
* performance status at least 80% according to Karnofsky scale and <2 according to WHO/ECOG scale
* cancer-related asymptomatic precachexia diagnosed
* absence of contraindications to oral nutrition and practicable realization of oral nutrition
* absence of severe, decompensated concomitant diseases
* signed informed consent for the participation in the study

Exclusion Criteria:

* diagnosis of a malignant neoplasm in clinical stage I-III
* disqualification from oncologic treatment
* cancer cachexia or cancer anorexia-cachexia syndrome
* poor performance status
* contraindications to oral nutrition or to high protein nutrition
* regular nutritional support at the moment of qualification to the study
* patient incompliance at the moment of qualification to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Chemotherapy-related toxicity during 12th week of observation | at baseline and after 12th week
  graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE Version 4.0); to determine whether nutritional support with high protein ONS in adult oncologic patients in the first step of cancer cachexia - asymptomatic precachexia, influence on the toxicity of systemic therapy during 3 months observation period (comparison of the results at the baseline and after 12 weeks)

SECONDARY OUTCOMES:
Changes in the Nutritional status / metabolic status | at baseline and after 12th week
  the assessment according to Nutritional Risk Screening 2002 (NRS 2002), Subjective Global Assessment (SGA), body mass, body mass index (BMI), VAS for appetite, albumin, prealbumin, triglycerides, total cholesterol, fasting blood glucose, C-reactive protein (CRP), ferritin, complete blood count.
  Body mass (in kg) will measure by the scales (Tanita BC 420). Hight ( in cm) measure by Stadiometer (Tanita)
  Body mass index calculation (BMI) on the basis of the following formula:
  BMI = body weight / height2 (kg/m2).
  VAS for appetite is 100-mm line where 0 mm means "I had no appetite at all" and 100 mm means "My appetite was very good".
  Laboratory parameters will measured by routine laboratory methods. All results will be compared between study groups (ONS vs without ONS) at the same time point (eg. baseline group ONS vs baseline group without ONS)
Changes in the Quality of life and patients well-being | at baseline and after 12th week
  FAACT-ESPEN score Version 4 (Functional Assessment of Anorexia/Cachexia Therapy questionnaire) is a measure of the quality of life and it is completed by a patient, it has a total of 42 questions. Patients mark 0 (none) - 4 (very much) for each question. This tool consists of five subscales: functional well-being (7 items), physical well-being (7 items), social/family well-being (7 items), emotional well-being (6 items) and other aspects, including appetite (13 items).
  The maximum score is 168. The lower the score, the lower overall quality of life.
Changes in the Performance status | at baseline and after 12th week
  To performance status assessment will be used Kornofsky scale and ECOG scale. The Karnofsky score allows to quantify the overall state and quality of life of a patient with neoplastic disease who qualifies to receive chemotherapy. The score has a range from 0 to 100, where 100 represents the ideal state and 0 - death.
  The Eastern Cooperative Oncology Group(ECOG) score runs from 0 to 5, with 0 denoting perfect health and 5 death.

CONTACTS AND LOCATIONS:
Overall Officials: Sylwia Malgorzewicz, MD, PhD, Principal Investigator — University Clinical Centre, Gdansk, Poland
Locations (1):
- University Clinical Centre, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Yes
publication in nutritional and oncological journals, presentation on the congresses

REFERENCES:
- [Derived] Zietarska M, Malgorzewicz S. Quality of Life of Colorectal Cancer Patients Treated with Chemotherapy. Nutrients. 2026 Jan 7;18(2):191. doi: 10.3390/nu18020191. PMID 41599804